CLINICAL TRIAL: NCT04454476
Title: Reversal of Preneoplastic Metaplasia in the Stomach With MEK Inhibitor Treatment
Brief Title: Reversal of Preneoplastic Metaplasia in the Stomach With MEK Inhibitor
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, James Goldenring, Principal Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 2049
Record Dates: First submitted 2020-06-24; First posted 2020-07-01 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer; Metaplasia; Stage I Gastric Cancer; Initial-onset Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms; Metaplasia | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Trametinib treatment (Experimental)
  Interventions: Drug: Trametinib treatment; Procedure: Endoscopy

INTERVENTIONS:
Drug: Trametinib treatment — 1 mg taken by mouth once a day for 14 days
Procedure: Endoscopy — A tiny camera on the end of a long, flexible tube will be used to examine the stomach and take biopsies.

SUMMARY:
This is a study of the safety and effectiveness of Trametinib treatment in patients who have received successful endoscopic submucosal resection of a Stage I gastric cancer.

DETAILED DESCRIPTION:
Objectives:

* To evaluate the efficacy of Trametinib in reversing metaplasia in participants with Stage 1 gastric cancer
* To evaluate the safety of Trametinibin in Stage I gastric cancer patients

ELIGIBILITY:
Inclusion Criteria:

Primary registration

* Person having intact stomach after treatment of early gastric cancer or gastric adenoma
* Person whose treated gastric cancer histological type is intestinal type.
* Person whose treated gastric cancer or gastric adenoma was curatively resected.
* Person who does not have symptoms of gastric cancer recurrence.
* Person who can declare agreement for enrollment by understanding the study and signing the informed consent document after hearing the explanation.
* Person who can visit the hospital in accordance with the schedule.

Secondary registration

* Person who has gastric atrophy at endoscopy.
* Person who does not have symptoms of gastric cancer recurrence by endoscopy.
* Person who has intestinal metaplasia in stomach, histologically confirmed in biopsy specimens taken under endoscopy within 8 weeks prior to taking MEK inhibitor, Trametinib.

Exclusion Criteria:

* Person whose treated gastric cancer was diffuse or signet ring cancer.
* Person whose treated gastric cancer or gastric adenoma was not curatively resected.
* Person who has the history of other malignant disease.
* Person who had a significant improvement in metaplasia after eradication therapy for Helicobacter pylori within one year.
* Person who had plan of eradication Helicobacter pylori in 1 year 9 months
* Person who has history of previous Trametinib or other MEK inhibitor use.
* Person who has history of hypersensitivity to excipients.
* Person who entered clinical trial and took investigational new drug within 12 weeks.
* Presence of active infection other than chronic gastritis.
* Cardiac conditions as follows:

  * Uncontrolled hypertension (BP>=150/95 mm Hg despite medical therapy)
  * Acute myocardial infection within 6 months prior to starting treatment
  * Uncontrolled Angina (Canadian Cardiovascular Society grade II-IV even after medication)
  * Symptomatic heart failure NYHA Class II-IV
  * <45% in the past
  * Severe valvular disease
  * <55% at present
  * Atrial fibrilation in ECG with BPM=>100 Laboratory values as listed below (SI units) Absolute Neutrophil Count <1.5x10A9/L (1500 per mm3) Platelets <100x10A9/L (100,000 per mm3) Hemoglobin<=9.0 g /dL Serum creatinine >1.5 X upper limit of normal (ULN) Serum bilirubin >1.5 x ULN AST or ALT > 2.5 x ULN

Ophthalmological conditions as follows:

Current or past history of retinal pigment epithelial detachment (RPED)/central serous retinopathy (CSR) or retinal vein occlusion Intraocular pressure (IOP) > 21 mmHg or uncontrolled glaucoma (irrespective of IOP)

Male or female patients of reproductive potential and, as judged by the investigator, are not employing an effective method of birth control and pregnant female.

Breast feeding female Have refractory nausea and vomiting , chronic gastrointestinal diseases (e.g . inflammatory bowel disease), or significant bowel resection that would adversely affect the absorption / bioavailability of the orally administered study medication.

Person who has history of hyperrefractory for Trametinib methyl sulfoxide Person who has pneumonia under chest X-ray. Have evidence of any other significant clinical disorder or laboratory finding that, as judgedby the investigator, makes it undesirable for the patient to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Trametinib in reversing metaplasia: changes in cell lineages | About 12 months
  The ability of Trametinib treatment to decrease the presence of metaplastic cell lineages in biopsies of the lining of the stomach, while also allowing the return of normal cell lineages (i.e. acid-secreting parietal cells). Cell lineages will be identified by immunostaining of tissue sections from biopsies.
Safety of Trametinib treatment: adverse events | About 12 weeks
  Assessment of side effects induced during or after treatment with Trametinib.

CONTACTS AND LOCATIONS:
Overall Officials: James Goldenring, MD, Principal Investigator — Vanderbilt Medical Center
Locations (3):
- Japan (3):
  - Nagasaki University Hospital, Nagasaki
  - Nihon University School of Medicine, Tokyo
  - University of Tokyo Medical Center, Tokyo

IPD SHARING:
Plan to Share IPD: No